CLINICAL TRIAL: NCT04735419
Title: Development of a Serocorrelate of Protection Against Invasive Group B Streptococcus Disease
Acronym: iGBS3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Medical Research Council (Other Government); University of Nottingham (Other); Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020.0176
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Streptococcus Agalactiae Infection
Keywords: Vaccine; Pregnancy; case control study; serocorrelate of protection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum Bacterial isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases are defined as infants who develop invasive GBS disease (iGBS disease= isolation of GBS from a normally sterile site, i.e. blood or CSF) in the first 90 days of life.
  Interventions: Other: No intervention
- Controls: Controls are defined as infants who are exposed to the same serotype of GBS at birth as the case - but who do not develop iGBS disease in the first 90 days of life.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A multicentre study to provide evidence that the relationship between an immune marker value (anti-GBS IgG concentration) and the probability of invasive GBS (iGBS) disease in infants less than 90 days of age is sufficiently strong that a vaccine able to induce an immune response will lead to a meaningful decrease in the probability of iGBS disease.

DETAILED DESCRIPTION:
Group B Streptococcus (GBS) is a bacterium (a bug) that causes serious infections in young infants across the world. In 2015 it was estimated that there were at least 319,000 infants under 3 months of age with GBS disease worldwide, resulting in 90,000 deaths and at least 10,000 children with long term disabilities. Around 20% of all pregnant women carry GBS in their vagina and bowel and babies are exposed to GBS bacteria around the time of birth. The options for prevention are currently limited to offering antibiotics during labour.

A vaccine that could be given to pregnant women has the greatest potential to benefit mothers and babies worldwide. There are vaccines currently being tested in clinical trials, including in pregnant women. The iGBS3 study aims to find out what levels of immunity (usually measured as antibody) a woman needs to pass to her baby to protect the baby from getting GBS disease. This will allow us to predict what antibody level a vaccine has to achieve to be effective and then to get those vaccines licensed and implemented as quickly as possible.

To do this, the study need to take a small sample of cord blood from a very large number of women just after delivering their baby. The study will need to follow around 180 000 babies in order to find at least 170 babies with GBS disease (of which 100 will have disease with the most common type) and compare their levels of antibody in cord blood with 300 healthy babies exposed to the same GBS type. To achieve this, SGUL will work with the Nottingham Clinical Trials Unit to embed this study in their existing GBS3 Trial, in which 80 hospitals across England, Scotland and Wales will be involved for 2 years.

Study Design iGBS3 is a large, multicentre, prospective, unmatched case control study in the UK designed to compare levels of antibody in cord blood in mothers whose infants develop GBS disease (iGBS) and colonised mothers whose infants do not develop GBS disease. To achieve this, the project aim to recruit at least 170 babies with GBS disease (of which 100 will have disease with the most common type) and 300 healthy babies exposed to the same GBS type. An exploratory substudy will look into levels of antibody in cord blood in mothers whose infants develop severe bacterial or viral infections caused by pathogens other than GBS.

Duration The overall duration of the project is planned for 36 months. This includes 2 months set-up, 12 months recruitment for Phase 1, 4 months for interval analysis, 12 months recruitment for Phase 2, 6 months for final retrieval of data, analysis and write-up.

Two phases

1. Phase 1 - cord blood collection and blood from an infant at time of GBS disease to establish the correlation between antibody at time of disease and cord blood
2. Phase 2 - if Phase 1 demonstrates that the correlation is strong, then in Phase 2 collection of blood from disease cases is required only; if Phase 2 shows a weak correlation, then in Phase 2 prospective collection of cord blood will continue.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

For iGBS disease case recruitment, an infant is not eligible unless a parent/person with parental responsibility gives informed consent For iGBS disease control recruitment, a mother is not eligible unless she gives informed consent.

Min Age: 0 Days | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women giving birth in maternity units in England, Scotland and Wales participating in the GBS3 study and their infants in the first 3 month of life
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlates objective | 36 months
  • To provide initial data on the relationship between antibody and iGBS disease risk by estimating the odds ratio of iGBS disease for antibody concentrations above various thresholds for STIII
Kinetics objective | 12 months
  • To determine whether antibody concentrations obtained at the time of disease (acute disease sample) can be used to predict cord antibody concentrations at birth in cases of iGBS STIII disease

SECONDARY OUTCOMES:
Correlates other than STIII | 36 months
  • To provide data on the relationship between antibody and iGBS disease risk by estimating the odds ratio of iGBS disease for antibody concentrations above various thresholds for serotypes other than STIII as well as all serotypes combined
Kinetics other than STIII | 12 months
  • To determine whether antibody concentrations obtained at the time of disease (acute disease sample) can be used to predict cord antibody concentrations in cases for serotypes others than STIII and to see if any declines differ by serotype
Controls objective | 36 months
  • To generate sufficient controls of women colonised with STIII and other serotypes

OTHER OUTCOMES:
Risk reduction objective | 36 months
  • To combine case-control study results (odds ratios and antibody RCD curves at different cut-offs) with other data on antibody distribution in the population and iGBS disease risk to determine absolute risk reduction. This could then be combined with vaccine immunologic trial data when available to allow prediction of vaccine efficacy (the decrease in probability of iGBS disease in infants of vaccinated compared to unvaccinated mothers).
Other pathogens sub-study | 36 months
  • To provide data on the relationship between antibody and infant infections caused by pathogens other than GBS

CONTACTS AND LOCATIONS:
Overall Officials: Paul Heath, Principal Investigator — St George's, University of London
Locations (1):
- St George's University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided